CLINICAL TRIAL: NCT06545084
Title: Evaluation of Periapical Healing Following Endodontic Microsurgery With Leukocyte and Platelet Rich Fibrin (L-PRF)
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 855857
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Leukocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Leukocyte and Platelet Rich Fibrin — Leukocyte Platelet Rich Fibrin (L-PRF) is a collection of growth factors rich in proinflammatory cells that promote healing after dental surgery. A L-PRF clot is obtained by collecting blood from the subject, similar to a phlebotomist drawing blood via venipuncture. The blood samples are spun in a centrifuge using the recommended settings by the manufacture(1). The resultant product has separated the red blood cells from the L-PRF clot which is placed back into the subject to promote healing of the surgical site.

SUMMARY:
The purpose of the study is to evaluate peri-radicular healing after root-end surgery using Leukocyte and Platelet Rich Fibrin. The study population includes patients diagnosed with persistent periapical pathology and scheduled for Endodontic Microsurgery at the University of Pennsylvania School of Dental Medicine, Department of Endodontics. Patients undergoing routine endodontic microsurgery and who meet the inclusion criteria will be given the opportunity to opt in to receive L-PRF in the osteotomy site to promote bone formation. Healing will be assessed radiographically and clinically at six, twelve, eighteen, and twenty-four months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study, including the follow-up visits.
3. Male or Female age >18 years old.
4. In good general health (ASA 2 or less) with no contraindications for Endodontic Microsurgery.
5. Persistent endodontic periapical pathology Class A, B, or C according to the Kim and Kratchman classification (5)
6. Intact coronal restorations with no evidence of leakage or caries under the restoration.

Exclusion Criteria:

1. Minors.
2. Suspected root fractures.
3. ASA classification 3 or greater.
4. Periapical pathology Class D, E, or F according to the Kim and Kratchman classification (5).
5. Patients with history of Oral or IV Bisphosphonate use.
6. Patients may be excluded if their treatment team do not believe Endodontic microsurgery and L-PRF graft is in the patient's best interests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dental Clinic population.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Peri-radicular Healing | 12 and 24 months
  Evaluate Peri-radicular healing after Endodontic Microsurgery with the use of autologous L-PRF plug.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No